CLINICAL TRIAL: NCT06760442
Title: Radiographic Evaluation of Crestal Bone Changes Following Equi-crestal Versus Subcrestal Implant Placement in Mandibular Posterior Augmented Ridge. A Randomized Controlled Clinical Trial.
Brief Title: Crestal Bone Changes Following Equi-crestal Versus Subcrestal Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Crestal Bone Changes
Record Dates: First submitted 2025-01-03; First posted 2025-01-06 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-01

CONDITIONS: Implant Therapy; Augmentation, Alveolar Ridge
Keywords: crestal bone level changes; subcrestal implant position; crestal implant position; augmented ridge; dental implants

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not know whether the implant is placed crestal or subcrestal Outcome assessor (primary and secondary outcomes) & biostatistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcrestal implant placement (Active Comparator): Delayed implant placement 2 mm subcrestally in missing mandibular posterior site.
  Interventions: Procedure: Subcrestal implant placement
- Crestal implant placement (Active Comparator): Delayed implant placement equicrestally in missing mandibular posterior site.
  Interventions: Procedure: Crestal implant placement

INTERVENTIONS:
Procedure: Subcrestal implant placement — Delayed implant placement 2 mm subcrestally in missing mandibular posterior site.
  Arms: Subcrestal implant placement
Procedure: Crestal implant placement — Delayed implant placement equicrestally in missing mandibular posterior site.
  Arms: Crestal implant placement

SUMMARY:
Statement of problem: The stability of peri-implant bone is a crucial factor for the long-term success of dental implants, where crestal bone plays a significant role in both the primary as well as the long- term implant stability. A bone loss of 1.5 mm during the first year of loading has been acceptable according to the early standards. However, more bone stability can be expected with the development in implant designs and surfaces over the past decades.

Aim of the study: the aim of this study is to radiographically assess the crestal bone changes following delayed implant placement in mandibular previously augmented posterior sites, comparing cases with equicrestal implant placement with subcrestal implant placement

DETAILED DESCRIPTION:
Statement of problem: The stability of peri-implant bone is a crucial factor for the long-term success of dental implants, where crestal bone plays a significant role in both the primary as well as the long- term implant stability. A bone loss of 1.5 mm during the first year of loading has been acceptable according to the early standards. However, more bone stability can be expected with the development in implant designs and surfaces over the past decades.

Aim of the study: the aim of this study is to radiographically assess the crestal bone changes following delayed implant placement in mandibular previously augmented posterior sites, comparing cases with equicrestal implant placement with subcrestal implant placement.

Materials and methods: This prospective, parallel, randomized controlled clinical trial will have 36 participants who need implant placement at the posterior mandibular area where they previously received horizontal bone augmentation. They will be randomly allocated into 2 groups, where group A (test) will receive dental implant placed subcrestally and group B (control) will receive implant placed equicrestally. Crestal bone loss will be assessed by periapical radiographs at implant placement (T0), 3 months (T3), 6 months (T6), 12 months (T12) and 18 months (T18) following implant placement. Keratinized tissue width, and soft tissue thickness will be measured clinically by periodontal probe at the same time points. Buccal bone changes will be evaluated at 18 months compared with the preoperative cone beam computed tomography by fusion module. Patient satisfaction will be recorded at the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 21 years.
* Patients having augmented (by 50/50 particulate xenograft and autogenous bone) edentulous posterior site with vertical bone height of > 10 mm in the mandible with a width of ridge ≥ 7 mm

  * Adequate Inter-arch space for implant placement
  * Favorable occlusion (no traumatic occlusion).
* Good oral hygiene.•Accepts 18 months follow-up period (cooperative patient)
* The patient provides informed consent.

Exclusion Criteria:

* Patients with inadequate bone volume and/ or quality
* Patients with remaining roots or with signs of acute infection related to the area of interest.
* Patients having systemic conditions that interfere with normal wound healing
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits .
* Smoker patients.
* Pregnant women.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Crestal bone changes | at baseline,3, 6 ,12 and 18 months
  Periapical digital radiographs to determine the amount of crestal bone lose in mm

SECONDARY OUTCOMES:
Keratinized tissue width | at baseline, 3,6,12 and 18 months
  Keratinized tissue width using periodontal probe in mm
Patient satisfaction | at baseline, 6 ,12 and 18 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: hani el nahas professor, Professor, Study Chair — Misr International University
Locations (1):
- Misr International University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No